CLINICAL TRIAL: NCT01008540
Title: Cytomegalovirus Resistance in Transplant Patients and Bone Marrow Recipients in the Prophylaxis Era, a French Multicentric Cohort Study
Brief Title: Prospective Multicentric Study of Cytomegalovirus Resistance in Transplant Patients and Bone Marrow Recipients
Acronym: PHRC CMV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: I06016
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cytomegalovirus
Keywords: cytomegalovirus; resistance; transplantation; Patient coming to an French transplantation center for solid organ or bone marrow transplant, with information and signed consent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: depistage — Virus isolation from urine, blood, or any suitable sample in case of CMV disease Resistance phenotype to antivirals UL97 and UL54 genes sequencing from blood, urines or any suitable samples for resistance mutations detection and polymorphism study

SUMMARY:
The investigators aim is to determine the incidence of cytomegalovirus resistance to antivirals in a cohort study. The patients are included at their first CMV active infection and are followed during two years thereafter. When criteria for suspected resistance are meet, blood and urine samples are collected for virus isolation and further resistance phenotype, and for resistance genotype determination. Results are compared with baseline samples. Clinical information such as treatment, immunosuppressive regimen and clinical evolution will be collected. Through this study, the investigators aim to organize a national network for the detection and identification of CMV resistant strains that will be useful when new therapeutics will be available.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic bone marrow transplant recipient or solid organ transplant recipient, included in the cohort at the time of its firs active CMV infection (ie biological signs of CMV replication (viremia, ADN or ARN aemia, Antigenaemiapp65….) with or without fever, or clinical end organ disease symptoms

Exclusion Criteria:

* Patient without medical care.policy,
* patient that did not signed the médical consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Resistance incidence in our patients with subgroup analysis, by organ and by the use of prophylaxis or preemptive treatment

SECONDARY OUTCOMES:
Strain diversity in baseline isolates and in resistant isolates Frequency of known resistance mutations Identification of new resistance-related mutations.

CONTACTS AND LOCATIONS:
Overall Officials: ALAIN Sophie, MD, Principal Investigator — University Hospital, Limoges
Locations (33):
- France (33):
  - Virologie, Amiens
  - Virologie, Angers
  - Virologie, Besançon
  - Virologie - Hôpital Avicenne, Bobigny
  - Virologie, Bordeaux
  - Virologie, Brest
  - Virologie, Caen
  - Virologie, Clermont-Ferrand
  - Virologie, Dijon
  - Virologie, Fort de France
  - Virologie, Grenoble
  - Virologie, Lille
  - Bactériologie Virologie, Limoges
  - Virologie, Lyon
  - Virologie, Montpellier
  - Virologie, Nancy
  - Virologie, Nantes
  - Virologie, Nîmes
  - Virologie - Hôpital BICHAT, Paris
  - Virologie - Hôpital La Pitié Salpétrière, Paris
  - Virologie - Hôpital LARIBOISIERE, Paris
  - Virologie - Hôpital NECKER, Paris
  - Virologie - Hôpital SAINT-LOUIS, Paris
  - Virologie, Poitiers
  - Virologie, Reims
  - Virologie, Rennes
  - Virologie, Rouen
  - Virologie, Saint-Etienne
  - Virologie, Strasbourg
  - Virologie, Suresne
  - Virologie, Toulouse
  - Virologie, Tours
  - Virologie - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Background] Andouard D, Mazeron MC, Ligat G, Couvreux A, Pouteil-Noble C, Cahen R, Yasdanpanah Y, Deering M, Viget N, Alain S, Hantz S. Contrasting effect of new HCMV pUL54 mutations on antiviral drug susceptibility: Benefits and limits of 3D analysis. Antiviral Res. 2016 May;129:115-119. doi: 10.1016/j.antiviral.2016.02.004. Epub 2016 Feb 10. PMID 26872863
- [Derived] Germi R, Mariette C, Alain S, Lupo J, Thiebaut A, Brion JP, Epaulard O, Saint Raymond C, Malvezzi P, Morand P. Success and failure of artesunate treatment in five transplant recipients with disease caused by drug-resistant cytomegalovirus. Antiviral Res. 2014 Jan;101:57-61. doi: 10.1016/j.antiviral.2013.10.014. Epub 2013 Nov 1. PMID 24184983
- [Derived] Hantz S, Garnier-Geoffroy F, Mazeron MC, Garrigue I, Merville P, Mengelle C, Rostaing L, Saint Marcoux F, Essig M, Rerolle JP, Cotin S, Germi R, Pillet S, Lebranchu Y, Turlure P, Alain S; French CMV Resistance Survey Study Group. Drug-resistant cytomegalovirus in transplant recipients: a French cohort study. J Antimicrob Chemother. 2010 Dec;65(12):2628-40. doi: 10.1093/jac/dkq368. Epub 2010 Oct 20. PMID 20961907